CLINICAL TRIAL: NCT04168671
Title: Continuous Laryngoscopy During Exercise Testing in Patients With Asthma
Brief Title: CLE During Exercise Testing in Asthma
Acronym: CLEtesting
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Coronavirus pandemia
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Paula Kauppi, MD, PhD, MD, PhD, Chief Specialist, Helsinki University Central Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HUS/886/2018
Record Dates: First submitted 2019-04-23; First posted 2019-11-19 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Larynx; Obstruction; Vocal Cord Dysfunction
MeSH Terms: conditions — Laryngeal Diseases; Bites and Stings; Vocal Cord Dysfunction

STUDY DESIGN:
Intervention Model Description: Asthma vs severe asthma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Asthma (Other): Asthma and symptomatic during exercise
  Interventions: Diagnostic Test: Continuous laryngoscopy during exercise test
- Severe asthma (Other): Severe asthma and symptomatic during exercise
  Interventions: Diagnostic Test: Continuous laryngoscopy during exercise test

INTERVENTIONS:
Diagnostic Test: Continuous laryngoscopy during exercise test — Continuous laryngoscopy during exercise test

SUMMARY:
The purpose is to assess visualize the level of laryngeal obstruction and vocal cord dysfunction and to obtain more information on causes for dyspnea in asthma and severe asthma and to assess safety of CLE in patients with asthma and with severe asthma. Patients are examined if symptomatic during exercise.

DETAILED DESCRIPTION:
* Questionnaires to assess breathlessness before the test.
* CLE on ergometer bicycle using any laryngoscopy setup
* Ergometry with spirometry tests with ECG, oxygen saturation, blood pressure, inspiratory and expiratory flow volume curves, bronchodilator after the exercise test
* Work load of 40W with 3 minutes intervals and increase by 40W in women. In men, work load of 50W with 3 minutes intervals and increase by 50W starting from 50W. In elderly and more severely disease work load of 30W with 3 minutes intervals and increase by 30W.
* Recording of dyspnoea, leg fatigue and chest discomfort
* Assessment of asthma by asthma control test, spirometry, exhaled NO measurements.
* Severe asthma group: physician-diagnosed asthma, moderate-high dose inhaled glucorticoid steroids and a second controller drug, exacerbations and per oral glucocorticoid steroid courses at least 2 in the past 12 months and/or 50% of the past 12 months on per oral glucocorticoidsteroids

ELIGIBILITY:
Inclusion Criteria:

* physician diagnosed asthma
* symptomatic during exercise

Exclusion Criteria:

* FEV1 <60%
* respiratory infection in the last 14 days
* asthma excacerbation in the last 14 days
* unstable cardiovascular disease
* bleeding disorder
* anticoagulant treatment (other than ASA)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Laryngeal obstruction | From immediately before (-5 minutes) before the exercise test, during the test up to 30 minutes
  Semi-quantitative visual estimation of laryngeal obstruction in test

SECONDARY OUTCOMES:
Safety of CLE in asthma (Incidence of test-emergent adverse events) | From immediately before (-10 minutes) before the exercise test, during the test up to 30 minutes
  Incidence of test-emergent adverse events: nasal bleeding or pain, panic attack, bronchial obstruction.
Exercise capacity in CLE in asthma | From 0 minutes before the exercise test and during the test up to 30 minutes
  Maximal work load in exercise test measured by W max 4 min
Dyspnea in CLE in asthma | From 0 minutes before the exercise test and during the test up to 30 minutes
  Assessment of patient reported dyspnea in maximal exercise measured by scale from 0 to 10 (Borg's scale) (0 no symptoms - 10 maximal dyspnea)
Exercise induced lung function changes | Immediately before test (0 minutes), and 10 minutes and 20 minutes after the test
  Change from baseline FEV1 after the test

CONTACTS AND LOCATIONS:
Overall Officials: Paula Kauppi, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lawlor C, Smithers CJ, Hamilton T, Baird C, Rahbar R, Choi S, Jennings R. Innovative management of severe tracheobronchomalacia using anterior and posterior tracheobronchopexy. Laryngoscope. 2020 Feb;130(2):E65-E74. doi: 10.1002/lary.27938. Epub 2019 Mar 25. PMID 30908672
- [Background] Bardin PG, Low K, Ruane L, Lau KK. Controversies and conundrums in vocal cord dysfunction. Lancet Respir Med. 2017 Jul;5(7):546-548. doi: 10.1016/S2213-2600(17)30221-7. No abstract available. PMID 28664856